CLINICAL TRIAL: NCT06105515
Title: Laparoscopic and Endoscopic Collaborative Surgery as Rescue-treatment for Advanced Gastric Cancer in Patients Unfit for Surgery - the LE-RACUS Pilot Clinical Study
Brief Title: Laparoscopic and Endoscopic Collaborative Surgery as Rescue-treatment for Advanced Gastric Cancer
Acronym: LE-RACUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ioannis Rouvelas, MD, PhD, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1298-9641
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
Keywords: Laparoscopic and endoscopic collaborative surgery; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): The group that will receive the active treatment
  Interventions: Procedure: Laparoscopic and Endoscopic Collaborative Surgery (LECS)

INTERVENTIONS:
Procedure: Laparoscopic and Endoscopic Collaborative Surgery (LECS) — Minimal invasive surgery in collaboration between endoscopy and laparoscopic surgery, to locally remove the tumor

SUMMARY:
The standard treatment for advanced gastric cancer without metastases is gastrectomy, where the whole stomach or a large proportion is removed surgically together with regional lymph nodes. Some patients cannot tolerate this invasive procedure because of old age or comorbidities. A tumor left in place can cause local symptoms such as bleeding or outlet obstruction. In this study, the investigators want to test the safety and feasibility of Laparoscopic and Endoscopic Collaborative Surgery (LECS) as a less invasive treatment option to locally remove gastric tumors without requiring extensive surgery in these frail patients. LECS is a minimally invasive surgical technique where the tumor margin is first marked from the inside with a gastroscope, followed by surgical removal of the lesion under endoscopic guidance.

DETAILED DESCRIPTION:
In patients with advanced gastric cancer (AGC), laparoscopic gastrectomy with lymph node dissection in combination with chemotherapy is the recommended treatment for cases with curative intent. However, some patients cannot tolerate such demanding treatment because of comorbidities or advanced age. If gastrectomy or palliative chemotherapy cannot be offered the only remaining alternative is best supportive care.

Patients with AGC that cannot receive definitive surgical or oncological treatment can develop complications such as bleeding from the primary tumor or gastric outlet obstruction. Such complications can be difficult to manage by endoscopic means, and significantly impact the patients' quality of life.

Laparoscopic and endoscopic collaborative surgery (LECS) was reported by Hiki et al in 2008 as a treatment for submucosal tumors. With this method, the endoscopist first performs mucosal incision around the tumor followed by laparoscopic removal of the tumor with endoscopic guidance.

In Japan, the current indication for LECS is gastrointestinal stromal cell tumors with a size of 2-5 cm. LECS has also been described in two case reports as palliative treatment for patients with AGC without being in a state to undergo gastrectomy. To the best of the investigators' knowledge, no prospective trial has studied LECS for this indication. Compared with gastrectomy, LECS is a very safe and much less invasive technique with few severe adverse events. If the tumor could be completely resected with LECS, the risk for bleeding and other tumor-related complications could be diminished which could significantly benefit the patients and improve their quality of life.

In this study, the investigators want to test the safety and feasibility of performing LECS for patients who are unfit for standard treatment with gastrectomy. The patients will be screened for inclusion through a multidisciplinary team meeting. If they meet the inclusion criteria they will be asked to participate in the study on an outpatient meeting with a member of the research team. If the patient agrees to participate and can sign an informed consent, they will be booked for a LECS procedure. After the operation is performed, the patient will meet the researcher again 4-6 weeks later and will be asked to fill in two QoL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* pT2-T4aN0M0 gastric carcinoma
* Borrmann type 1-2 < 5 cm or Borrmann type 3 < 2 cm
* Patient assessment by the multidisciplinary tumor board as not fit for gastrectomy
* Signed informed consent

Exclusion Criteria:

* Borrman type 4
* Location in the cardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Severe complication | Through study completion, an average of 2 years
  Clavien Dindo complication grade >/= III

SECONDARY OUTCOMES:
Any complication | Through study completion, an average of 2 years
  Clavien Dindo complication grade II-IV
Postoperative bleeding/leakage/postoperative abcess | Through study completion, an average of 2 years
  Use of blood transfusion/abcess requiring drainage
Operation time/local radicality | Through study completion, an average of 2 years
  Time of the surgical procedure/pathology report of radical resection
30-day mortality/in-hospital mortality/hospital-stay | Through study completion, an average of 2 years
  Mortality within 30 days/mortality during the hospital stay/number of days admitted
Health-related quality of life | Through study completion, an average of 2 years
  The QLQ-C30/OG25 HQL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Rouvelas, MD, PhD, Principal Investigator — ME Övre buk, Karolinska Universitetssjukhuset
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Yu F, Wu L, Ye F, Zhang L, Li Y. Survival after Gastrectomy in Node-Negative Gastric Cancer: A Review and Meta-Analysis of Prognostic Factors. Med Sci Monit. 2015 Jul 2;21:1911-9. doi: 10.12659/MSM.893856. PMID 26134762
- [Background] Hiki N, Yamamoto Y, Fukunaga T, Yamaguchi T, Nunobe S, Tokunaga M, Miki A, Ohyama S, Seto Y. Laparoscopic and endoscopic cooperative surgery for gastrointestinal stromal tumor dissection. Surg Endosc. 2008 Jul;22(7):1729-35. doi: 10.1007/s00464-007-9696-8. Epub 2007 Dec 12. PMID 18074180
- [Background] Takechi H, Fujikuni N, Takemoto Y, Tanabe K, Amano H, Noriyuki T, Nakahara M. Palliative surgery for advanced gastric cancer: Partial gastrectomy using the inverted laparoscopic and endoscopic cooperative surgery method. Int J Surg Case Rep. 2018;50:42-45. doi: 10.1016/j.ijscr.2018.06.042. Epub 2018 Jul 21. PMID 30077165
- [Background] Washio M, Hiki N, Hosoda K, Niihara M, Chuman M, Sakuraya M, Wada T, Harada H, Sato T, Tanaka K, Naitoh T, Kumamoto Y, Sangai T, Tanabe S, Yamashita K. Laparoscopic and endoscopic cooperative surgery for advanced gastric cancer as palliative surgery in elderly patients: a case report. Surg Case Rep. 2021 Nov 15;7(1):241. doi: 10.1186/s40792-021-01325-1. PMID 34779942
- [Background] de Brito SO, Libanio D, Pinto CMM, de Araujo Teixeira JPPO, de Araujo Teixeira JPM. Efficacy and Safety of Laparoscopic Endoscopic Cooperative Surgery in Upper Gastrointestinal Lesions: A Systematic Review and Meta-Analysis. GE Port J Gastroenterol. 2022 Nov 7;30(1):4-19. doi: 10.1159/000526644. eCollection 2023 Jan. PMID 36743984
- [Derived] Maltzman H, Omae M, Klevebro F, Baldaque-Silva F, Rouvelas I. Laparoscopic and Endoscopic cooperative surgery as Rescue-treatment for Advanced gastric Cancer in patients Unfit for Surgery (LE-RACUS): protocol for a feasibility study. Pilot Feasibility Stud. 2025 Jan 3;11(1):1. doi: 10.1186/s40814-024-01584-3. PMID 39754254